CLINICAL TRIAL: NCT06375083
Title: Implementing Computerized Cognitive Behavioral Therapies for Suicide Prevention and Depression Among At-Risk Rural and Urban Veterans
Brief Title: Computerized Cognitive Behavioral Therapies for Suicide Prevention and Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-1231
Record Dates: First submitted 2023-09-19; First posted 2024-04-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Suicide; Depression
Keywords: Suicide; Depression; Veterans; Cognitive Behavioral Therapy
MeSH Terms: conditions — Suicide; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Cognitive Behavioral Therapy for Suicide Prevention (cCBT-SP) and Cognitive Behavioral Therapy for Depression (cCBT-D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Online (computerized) CBT for Depression or Suicide Prevention
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The computerized Cognitive Behavioral Therapy for Suicide Prevention (cCBT-SP) course is comprised of 12 online sessions and is augmented by use of a companion workbook. The computerized Cognitive Behavioral Therapy for Depression (cCBT-D) course is comprised of 12 online sessions.

SUMMARY:
This study plans to learn more about the use of one of two self-guided online cognitive behavioral therapy courses. One is focused on symptoms of depression and one is focused on history of suicidal thoughts and behaviors.

DETAILED DESCRIPTION:
Based on previous work with other computerized CBT (cCBT) interventions (e.g., cCBT-D), which has found that cCBT has similar effectiveness to traditional CBT, members of the team along with Veterans Health Administration (VHA) leaders have developed computerized cCBT-SP and cCBT-D courses that will be ready for safety, feasibility, and acceptability testing. If proven to be feasible, safe, and effective, these courses could be made available to all Veterans, at no cost to users.

ELIGIBILITY:
Cohort A - cCBT-SP Program

Inclusion Criteria:

1. Veterans between the ages of 18 and 65
2. Currently living in Colorado, New York, Montana, Texas, or Utah who have accessed VA Care
3. Recent suicidal ideation (past month; C-SSRS Screener -Yes to Item 2) and history of lifetime suicidal behavior (lifetime, C-SSRS Screener - Yes to Item 6)
4. Reliable access to a computer/tablet and the internet
5. Ability to provide informed consent

Exclusion Criteria:

1. Active alcohol or substance use disorder, excluding Cannabis dependence, as determined by screening or electronic medical record
2. Identification of active psychosis or bipolar disorder, as determined via screening or electronic medical record
3. Severe cognitive impairment, as determined by screening or electronic medical record
4. Currently enrolled in/participating in another mental health-related intervention research study

Cohort B - cCBT-D Program

Inclusion Criteria:

1. Veterans between the ages of 18 and 65
2. Currently living in Colorado, New York, Montana, Texas, or Utah who have accessed VA care
3. Mild to moderate depressive symptoms, as determined by the PHQ-9, (score of 5-14)
4. Reliable access to a computer/tablet and the internet
5. Ability to provide informed consent

Exclusion Criteria:

1. PHQ-9 score below 4 or 15 and above
2. Active alcohol or substance use disorder, excluding Cannabis dependence, as determined by screening or electronic medical record
3. Identification of active psychosis or bipolar disorder, as determined via screening or electronic medical record
4. Severe cognitive impairment, as determined by screening or electronic medical record
5. Currently enrolled in/participating in other intervention research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 12 weeks
  Acceptability
Internet Evaluation and Utility Questionnaire | 12 weeks
  Acceptability
Internet Impact and Effectiveness Questionnaire | 12 weeks
  Acceptability
Narrative Evaluation of Intervention Interview | 12 weeks
  Acceptability
Recruitment Rate | 12 weeks
  Number of individuals who consented to participate
Completion of intervention | 12 weeks
  Number of participants who completed most or all of the sessions

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation | 12 weeks
  Change in suicidal ideation
Patient Health Questionnaire-9 | 12 weeks
  Change in depression symptoms
Posttraumatic Stress Disorder Checklist-5 | 12 weeks
  Change in PTSD symptoms
Generalized Anxiety Disorder-7 | 12 weeks
  Change in anxiety symptoms
Computerized Adaptive Testing - Suicide Scale | 12 weeks
  Change in suicidal ideation

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- Eastern Colorado Health Care System, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No